CLINICAL TRIAL: NCT00182884
Title: Preventing Delirium in Hospitalized Elderly
Brief Title: Donepezil in Preventing Delirium in Hospitalized Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University Health (Other)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IA0079; VFR-161
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2008-02

CONDITIONS: Postoperative Complications; Delirium
Keywords: Hospital acquired complications; adverse effects; Cognitive Impairment; Aging
MeSH Terms: conditions — Postoperative Complications; Delirium; Cognitive Dysfunction | interventions — Donepezil

INTERVENTIONS:
Drug: Donepezil

SUMMARY:
The purpose of this study is to explore the efficacy of a perioperative daily dose of Donepezil (a cholinergic enhancer) in reducing the incidence and severity of delirium.

DETAILED DESCRIPTION:
Delirium is confusion or a sudden change in alertness which may happen after hip repair surgery. Up to 65% of elderly undergoing surgical repair of hip fracture experience post-operative delirium. These individuals often stay in the hospital longer, have more complications, and are more likely to die. Early studies suggest that delirium could be prevented by correcting the central cholinergic deficit that is associated with delirium. Donepezil is currently being used to treat memory loss in patients with Alzheimer's disease.

This study will recruit 30 adults aged 65 or older who are undergoing hip fracture surgery. Participants will be randomized to receive either Donepezil or a matching placebo within 24 hours prior to surgery and for 4 days after the surgery.

All material to be collected will be from interviews, questionnaires, and medical chart review at baseline and daily for the entire hospital stay. The Confusion Assessment Method (CAM) and Memorial Delirium Assessment Scale (MDAS) will be used to evaluate the effect of Donepezil on delirium incidence and severity. Other assessments include cognitive deficit, length of hospitalization, discharge site, adverse effects, and psychotropic medications.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling individuals aged 65 or older
* Admitted to Methodist Hospital for surgical repair of hip fracture
* No evidence of delirium at admission to hospital
* MMSE total score below 24 points after adjustment for education and age
* Consent to participate in the study

Exclusion Criteria:

* Severely demented as defined by MMSE score below 10
* Metastatic cancer or other comorbid illnesses likely to reduce life expectancy to under 6 months
* Multiple trauma or pathological fractures
* Aphasic, legally blind, or deaf
* Use of Donepezil or other cholinesterase inhibitors within one month prior to surgery
* Allergy to Donepezil

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30
Dates: Start 2004-07; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Postoperative cumulative incident cases of delirium, as defined by the Confusion Assessment Method (CAM) administered at baseline prior to surgery and daily until discharge
delirium severity as measured by the Memorial Delirium Assessment Scale (MDAS)

SECONDARY OUTCOMES:
Cognitive status as measured by the Mini Mental Status Exam (MMSE)
behavioral status using the Rating Scale for Aggressive Behavior in the Elderly (RAGE)
length of stay in hospital postoperatively
discharge site
adverse effects
use of psychotropic medications

CONTACTS AND LOCATIONS:
Overall Officials: Malaz Boustani, MD, MPH, Principal Investigator — Regenstrief Institute, Indiana University Center for Aging Research
Locations (1):
- Methodist Hospital, Clarian Health Partners, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Cooper C, Campion G, Melton LJ 3rd. Hip fractures in the elderly: a world-wide projection. Osteoporos Int. 1992 Nov;2(6):285-9. doi: 10.1007/BF01623184. PMID 1421796
- [Background] Cummings SR, Rubin SM, Black D. The future of hip fractures in the United States. Numbers, costs, and potential effects of postmenopausal estrogen. Clin Orthop Relat Res. 1990 Mar;(252):163-6. PMID 2302881
- [Background] Barrett-Connor E. The economic and human costs of osteoporotic fracture. Am J Med. 1995 Feb 27;98(2A):3S-8S. doi: 10.1016/s0002-9343(05)80037-3. No abstract available. PMID 7709931
- [Background] Galanakis P, Bickel H, Gradinger R, Von Gumppenberg S, Forstl H. Acute confusional state in the elderly following hip surgery: incidence, risk factors and complications. Int J Geriatr Psychiatry. 2001 Apr;16(4):349-55. doi: 10.1002/gps.327. PMID 11333420
- [Background] Gustafson Y, Berggren D, Brannstrom B, Bucht G, Norberg A, Hansson LI, Winblad B. Acute confusional states in elderly patients treated for femoral neck fracture. J Am Geriatr Soc. 1988 Jun;36(6):525-30. doi: 10.1111/j.1532-5415.1988.tb04023.x. PMID 2897391